CLINICAL TRIAL: NCT02777151
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study Investigating the Safety, Tolerability, and Pharmacokinetics of Intravenously Administered REGN3470-3471-3479 in Healthy Adult Subjects
Brief Title: Study of Safety, Tolerability, and Pharmacokinetics of REGN3470-3471-3479 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R3470-3471-3479-HV-1528
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — atoltivimab, maftivimab, and odesivimab-ebgn drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): REGN3470-3471-3479 dosing level 1 or placebo
  Interventions: Drug: REGN3470-3471-3479; Drug: Placebo
- Cohort 2 (Experimental): REGN3470-3471-3479 dosing level 2 or placebo
  Interventions: Drug: REGN3470-3471-3479; Drug: Placebo
- Cohort 3 (Experimental): REGN3470-3471-3479 dosing level 3 or placebo
  Interventions: Drug: REGN3470-3471-3479; Drug: Placebo
- Cohort 4 (Experimental): REGN3470-3471-3479 dosing level 4 or placebo
  Interventions: Drug: REGN3470-3471-3479; Drug: Placebo

INTERVENTIONS:
Drug: REGN3470-3471-3479
Drug: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, dose escalation study evaluating the safety, tolerability, pharmacokinetics (PK) and immunogenicity of REGN3470-3471-3479 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man or woman between the ages of 18 and 60
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent
5. Able to understand and complete study-related questionnaires

Exclusion Criteria:

1. Use of any medications started within 30 days prior to the screening visit including, prescription medications, nutritional supplements, and over-the-counter medications except for vitamin supplements, and recommended doses of acetaminophen, aspirin or ibuprofen
2. Hospitalization for any reason within 60 days prior to the screening visit
3. History of or positive human immunodeficiency virus (HIV) screen result at the screening visit
4. History of or positive blood test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) or hepatitis C virus (HCV) antibody at the screening visit
5. History of drug or alcohol abuse within 1 year prior to screening
6. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit
7. Any history of receiving treatment, vaccine or mAbs against the Ebola virus
8. Pregnant or breast-feeding women
9. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

   * Contraception is not required for men with documented vasectomy.
   * Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. A baseline follicle-stimulating hormone (FSH) test will be performed for confirmation of menopausal status. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs through the end of the study visit in subjects treated with REGN3470-3471-3479 in a fixed dose combination | From baseline up to day 169

SECONDARY OUTCOMES:
Concentration of REGN3479 in serum over time | From baseline up to day 169
Concentration of REGN3471 in serum over time | From baseline up to day 169
Concentration of REGN3470 in serum over time | From baseline up to day 169
The presence or absence of antibodies against REGN3470 over time | From baseline up to day 169
The presence or absence of antibodies against REGN3471 over time | From baseline up to day 169
The presence or absence of antibodies against REGN3479 over time | From baseline up to day 169

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sivapalasingam S, Kamal M, Slim R, Hosain R, Shao W, Stoltz R, Yen J, Pologe LG, Cao Y, Partridge M, Sumner G, Lipsich L. Safety, pharmacokinetics, and immunogenicity of a co-formulated cocktail of three human monoclonal antibodies targeting Ebola virus glycoprotein in healthy adults: a randomised, first-in-human phase 1 study. Lancet Infect Dis. 2018 Aug;18(8):884-893. doi: 10.1016/S1473-3099(18)30397-9. Epub 2018 Jun 18. PMID 29929783